CLINICAL TRIAL: NCT02183519
Title: Respiratory Kinematics of Reflex and Voluntary Cough in Healthy Older Adults and Parkinson's Disease
Brief Title: Respiratory Kinematics of Cough in Healthy Older Adults and Parkinson's Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB201400477
Record Dates: First submitted 2014-07-02; First posted 2014-07-08 (Estimated); Results first posted 2017-03-24 (Actual); Last update posted 2017-03-24 (Actual); Status verified 2017-02

CONDITIONS: Cough; Parkinson's Disease
Keywords: Cough; Reflex; Voluntary; Healthy older adults; Parkinson's disease; Respiratory kinematics; Cueing
MeSH Terms: conditions — Cough; Parkinson Disease | interventions — Capsaicin

STUDY DESIGN:
Intervention Model Description: Participants with Parkinson's Disease are evaluated in parallel against a control group of health older adults
Masking Description: 1) baseline respiratory maneuvers for calibration of the Respitrace system with spirometry 2) sequential voluntary cough (no cueing), 3) reflex cough sensitivity testing to establish the lowest concentration of capsaicin that elicits a two cough response (C2) (no cueing), 4) randomized production of sequential voluntary cough (3x) or reflex cough induced with C2 (3x) with cueing to 'cough long and hard' and 5) flexible laryngoscopy to assess age-related changes to the larynx that may impact cough function.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Healthy older adults (Experimental): All participants will receive reflex and voluntary cough testing. This will include coughing on command (voluntary cough) and coughing in response to capsaicin (reflex cough). This data will me measured to determine the strength of the cough (from both voluntary and reflex cough) and cough sensitivity (reflex cough only). Following baseline reflex and voluntary cough assessment, the participants will be cued to cough long and hard during both reflex and voluntary cough tasks. These data will help the investigators understand the baseline characteristics of voluntary and reflex cough, whether older adults can modify the magnitude of their cough response with verbal and visual cues.
  Interventions: Drug: Capsaicin; Other: Voluntary cough test
- Parkinson's disease (Experimental): All participants will receive reflex and voluntary cough testing. This will include coughing on command (voluntary cough) and coughing in response to capsaicin (reflex cough). This data will me measured to determine the strength of the cough (from both voluntary and reflex cough) and cough sensitivity (reflex cough only). Following baseline reflex and voluntary cough assessment, the participants will be cued to cough long and hard during both reflex and voluntary cough tasks. These data will help the investigators understand the baseline characteristics of voluntary and reflex cough, whether older adults can modify the magnitude of their cough response with verbal and visual cues.
  Interventions: Drug: Capsaicin; Other: Voluntary cough test

INTERVENTIONS:
Drug: Capsaicin — For reflex cough testing, all participants will receive various concentrations of nebulized capsaicin. Delivery of multiple concentrations and doses of capsaicin allows for accurate assessment of both the strength (airflow measures) of reflex, as well as cough sensitivity.
Other: Voluntary cough test — Participants will be fitted with a facemask covering their mouth and nose, and instructed to cough into the facemask.

SUMMARY:
The purpose of this research study is to test cough function in individuals with Parkinson's disease and healthy older adults. Cough is a complex, defensive function which involves movement of the chest and lungs. The investigators want to compare the movement of the chest wall and the lungs during voluntary and reflex cough.

The long-term goal of this research is to develop treatments for people with cough dysfunction. Cough dysfunction increases the risk for respiratory infections such as pneumonia. The results from this study will provide information to help researchers understand the difference between reflex and voluntary cough more fully.

DETAILED DESCRIPTION:
If the participant agrees to participate, the investigators will first test pulmonary (lung) function. Next, the investigators will test voluntary and reflex cough. After this first round of cough testing, the investigators will ask participants to cough long and hard during voluntary and reflex cough testing. Finally, the investigators will view the larynx (voice box) with an endoscopic camera inserted through the nose. This test is done to see if there are any changes in the larynx that may influence cough.

ELIGIBILITY:
Inclusion Criteria:

* Age 55-85 years
* Ability to provide informed consent

For participants with Parkinson's disease (PD):

- Diagnosis of PD (Hoehn & Yahr stages II-IV) by a University of Florida Movement Disorders fellowship trained neurologist having completed a clinical assessment of each participant's PD severity and arriving at the diagnosis of PD by applying strict United Kingdom brain bank criteria.

Exclusion Criteria:

Participants with PD:

- History of neurological disorders other than PD (e.g. multiple sclerosis, stroke, brain tumor, etc)

Healthy older adults:

* History of neurological disease including PD
* History of head and neck cancer
* History of breathing disorders or disease (i.e. chronic obstructive pulmonary disease, asthma)
* History of smoking for more than 5 years at any one time (as this reduces the sensitivity to capsaicin)
* History of chest infection the last 5 weeks
* Failure of a screening test of pulmonary function (e.g. forced expiratory volume in one second/forced vital capacity<75%)
* Difficulty complying due to neuropsychological dysfunction (i.e. severe depression)

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2014-10; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen W. Hegland, Ph.D., Principal Investigator — University of Florida; Alexandra E. Brandimore, M.A. CCC/SLP, Study Director — University of Florida
Locations (2):
- United States (2):
  - Center for Movement Disorders and Neurorestoration, Gainesville, Florida
  - Dauer Hall, University of Florida, Gainesville, Florida

REFERENCES:
- [Background] Smith JA, Aliverti A, Quaranta M, McGuinness K, Kelsall A, Earis J, Calverley PM. Chest wall dynamics during voluntary and induced cough in healthy volunteers. J Physiol. 2012 Feb 1;590(3):563-74. doi: 10.1113/jphysiol.2011.213157. Epub 2011 Dec 5. PMID 22144580

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Parkinson's Disease = PD and Healthy Older Adult = HOA
Pre-assignment Details: 10 PD participants did not respond to 200micro-molar capsaicin, and received the 500 micro-molar single dose. 3/10 PD participants did not respond to 500, and thus did not produce analyzable data. Due to a computer error, data was lost for 3 of the HOA participants. Complete data sets were analyzed for 13 PD and 25 HOA participants.
Period: Overall Study
Arm/Group | Healthy Older Adults | Parkinson's Disease
Started | 28 | 16
Completed | 25 | 13
Not Completed | 3 | 3
Not completed — computer error | 3 | 0
Not completed — Did not respond to cough inducter | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Older Adults | Parkinson's Disease | Total
Number analyzed (Participants) | 25 | 13 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 2 | 7
  >=65 years | 20 | 11 | 31
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 6 | 17
  Male | 14 | 7 | 21
Region of Enrollment [Number; unit: participants]
  United States | 25 | 13 | 38

OUTCOME MEASURES:

1. Primary Outcome: Peak Expiratory Flow Rate
Description: Peak expiratory flow rate is the maximum volume of air that is expelled per unit time for each cough in a cough epoch. Measured in liters/second.
Time Frame: 1-2 hours
Measure: Mean (Standard Deviation); unit: Liters of air/second
Arm/Group | Healthy Older Adults | Parkinson's Disease
Number analyzed (Participants) | 25 | 13
Liters of air/second | 4.34 (.202) | 3.92 (.274)

ADVERSE EVENTS:
Arm/Group | Healthy Older Adults | Parkinson's Disease
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/13
Other Adverse Events (participants affected / at risk) | 0/25 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes